CLINICAL TRIAL: NCT00001541
Title: Analysis of Bronchial and Bronchoalveolar Lavage Fluid and Bronchial Mucosal Biopsies in Patients With Wegener's Granulomatosis
Brief Title: Analysis of Bronchial Tissue and Fluid in Patients With Wegener's Granulomatosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960065; 96-I-0065
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-01

CONDITIONS: Inflammation; Vasculitis; Wegener's Granulomatosis
Keywords: Vasculitis; Inflammation; Bronchoscopy; Cytokines; Inflammatory Mediators; Wegener's Granulomatosis
MeSH Terms: conditions — Inflammation; Vasculitis; Granulomatosis with Polyangiitis

SUMMARY:
This study will collect fluid and tissue samples from the bronchi (air passages to the lungs) of patients with Wegener's granulomatosis for laboratory examination. Wegener's granulomatosis is a type of vasculitis (blood vessel inflammation) that can affect many parts of the body, including the brain, nerves, eyes, skin, sinuses, kidneys, intestinal tract, joints, heart, lungs and other sites. About 85 percent of patients have lung involvement. The lining of the bronchi (bronchial mucosa) is composed of cells that produce mucus, inflammatory cells, and inflammatory mediators (chemicals produced in response to inflammation). Analysis of these various substances may provide insight into what causes different types of lung problems in Wegener's granulomatosis.

Patients between 18 and 75 years of age with Wegener's granulomatosis who require bronchoscopy to evaluate the cause of their lung problem may be eligible for this study.

Participants will undergo a bronchoscopy in the hospital intensive care unit (ICU). For this procedure, the mouth and throat are numbed with lidocaine jelly and spray. If needed, a sedative is given for comfort. A small plastic tube (intravenous catheter) is placed in a vein to give medications. A pencil-thin tube is then placed through the nose or mouth into the lung airways to examine the airways carefully.

At the time of the bronchoscopy, patients in this study will undergo the following additional procedures:

* Bronchoalveolar lavage - Saline (salt water) is injected through the bronchoscope into the air passage, acting as a rinse. A sample of the fluid is then withdrawn and examined for infection, inflammatory cells and inflammatory chemicals. (This may be done as part of the standard medical care procedure.)
* Bronchial lavage - This procedure is similar to bronchoalveolar lavage, but less fluid is used to rinse larger airways.
* Bronchial mucosal biopsies - A small wire is inserted through the bronchoscope next to the bronchial lining. Forceps at the end of the wire pinch off a small piece of tissue for withdrawal and examination.

The patient's heart rhythm and rate and oxygen levels are monitored during the procedure. When the procedures are finished, the patient is monitored in the ICU until the numbing effect of the anesthetic has worn off and then moves to a regular hospital bed for overnight.

Patients whose test results show an isolated infection or isolated Wegener's lung tissue involvement and who are being treated or are eligible for treatment under another NIH protocol will be followed by X-ray for improvement of their infection or other lung involvement with treatment. Patients whose infection or lung tissue involvement improves may be asked to undergo a second bronchoscopy as described above, but for research purposes only.

DETAILED DESCRIPTION:
Wegener's granulomatosis is a systemic vasculitis in which parenchymal and/or endobronchial inflammation frequently occur. The purpose of this investigation is to analyze bronchial and bronchoalveolar lavage fluid in patients with Wegener's granulomatosis for the presence of immunoregulatory mediators and pro-inflammatory cytokines. We will also be examining mucosal biopsies in these patients to define the histologic changes, the phenotype of infiltrating leukocytes, and the pattern of adhesion molecule expression that may be present. Such studies could lead to an improved understanding of the pathophysiology of this disease and of its pulmonary manifestations and provide potential directions for future therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

Diagnosis of Wegener's granulomatosis based on clinical and histological characteristics.

Age between 18-75 years.

Bronchoscopy is required as part of their standard medical care.

FEV1 is greater than 55 percent of FVC.

O2 saturation is greater than 90 percent.

EXCLUSION CRITERIA:

FEV1 is less than 55% of FVC.

O2 saturation is less than 90%.

Abnormal PT, PTT, or platelet count less than 50.

History of adverse reaction to lidocaine or other local anesthetics.

Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1996-04; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Levine SJ. Bronchial epithelial cell-cytokine interactions in airway inflammation. J Investig Med. 1995 Jun;43(3):241-9. PMID 7614070
- [Background] Shelhamer JH, Levine SJ, Wu T, Jacoby DB, Kaliner MA, Rennard SI. NIH conference. Airway inflammation. Ann Intern Med. 1995 Aug 15;123(4):288-304. doi: 10.7326/0003-4819-123-4-199508150-00008. PMID 7611596
- [Background] Hoffman GS, Sechler JM, Gallin JI, Shelhamer JH, Suffredini A, Ognibene FP, Baltaro RJ, Fleisher TA, Leavitt RY, Travis WD, et al. Bronchoalveolar lavage analysis in Wegener's granulomatosis. A method to study disease pathogenesis. Am Rev Respir Dis. 1991 Feb;143(2):401-7. doi: 10.1164/ajrccm/143.2.401. PMID 1990960